CLINICAL TRIAL: NCT03268603
Title: A Phase II Study of Intrathecal Autologous Adipose-derived Mesenchymal Stromal Cells for Amyotrophic Lateral Sclerosis
Brief Title: Intrathecal Autologous Adipose-derived Mesenchymal Stromal Cells for Amyotrophic Lateral Sclerosis (ALS)
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: State of Minnesota Regenerative Medicine Minnesota (Unknown)
Responsible Party: Principal Investigator, Nathan P. Staff, Professor of Neurology, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 15-008008
Record Dates: First submitted 2017-08-30; First posted 2017-08-31 (Actual); Results first posted 2025-04-02 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: ALS; Amyotrophic Lateral Sclerosis
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Mesenchymal Stromal Cells (Experimental): Autologous Adipose-derived Mesenchymal Stromal Cells (aaMSCs) will be administered intrathecally at a single dose in a volume of 5-10 mL, all patients will receive 5 x 10^7 intrathecal aaMSCs at the first injection (Visit 4). Subsequent doses may be reduced to 1 x 10^7 or increased to 1 x 10^8, based on Dose Modification Rules.
  Interventions: Drug: Autologous Adipose-derived Mesenchymal Stromal Cells

INTERVENTIONS:
Drug: Autologous Adipose-derived Mesenchymal Stromal Cells — The investigational product consists of autologous adipose-derived Mesenchymal Stromal Cells (MSCs), suspended in 5-10 mL Lactated Ringer's. The MSC are provided in a sterile syringe labelled with appropriate patient and product identifiers ready for intrathecal injection.

SUMMARY:
The purpose of this study is to determine the safety and efficacy of intrathecal treatment delivered to the cerebrospinal fluid (CSF) of mesenchymal stem cells in ALS patients every 3 months for a total of 4 injections over 12 months.

Mesenchymal stem cells (MSCs) are a type of stem cell that can be grown into a number of different kinds of cells. In this study, MSCs will be taken from the subject's body fat and grown. CSF is the fluid surrounding the spine.

The use of mesenchymal stem cells is considered investigational, which means it has not been approved by the Food and Drug Administration (FDA) for routine clinical use. However, the FDA has allowed the use of mesenchymal stem cells in this research study.

DETAILED DESCRIPTION:
The Goal of the Proposed Study is to perform an open label, 60 subject, Phase II multi-site clinical trial to investigate the safety and efficacy of intrathecal treatment of aaMSCs in ALS. Patients will be treated with 10-100 million aaMSCs every 3 months for a total of 4 intrathecal injections over 12 months. Reduced dose treatments will be allowed based on specific adverse events. Multiple biomarkers will be tracked throughout the clinical trial and correlated with response to treatment. This study was initially performed at Mayo Clinic in Rochester and subsequently expanded to the two other Mayo Clinic sites in Arizona and Florida. All biopsies and stem cell injections take place at Mayo Clinic Rochester, regardless of where the subject initially enrolls into the study.

ELIGIBILITY:
Inclusion Criteria:

* All patients will have ALS diagnosed as possible, laboratory-supported probable, probable, or definite as defined by the World Federation of Neurology criteria for the diagnosis of ALS.
* Examination and neurophysiological testing confirm a pure motor syndrome compatible with the diagnosis of ALS. All other possible causes of weakness have been excluded by extensive investigations.
* Age greater than 18 years, if female, must be post-menopausal, had a hysterectomy, or agree to two forms of birth control.
* Permanent resident or citizen of the United States.
* Geographic accessibility to the study site and willingness and ability to comply with follow-up.
* History of a chronic onset of a progressive motor weakness of less than two years duration.
* Subjects must be taking a stable dose of riluzole for at least 30 days prior to enrolment or not be on riluzole, and not have been on it for at least 30 days prior to enrolment (riluzole-naïve subjects are permitted in the study).
* Subjects must be taking a stable dose of oral Radicava® (edaravone) for at least 30 days prior to enrolment or not be on oral Radicava® (edaravone), and not have been on it for at least 30 days prior to enrolment (edaravone-naïve subjects are permitted in the study).
* Able to comply with protocol requirements, including MRI testing.
* Can provide written informed consent.

Exclusion Criteria:

* Use of Radicava® (edaravone) within 30 days of screening or intent to use Radicava® at any time during the course of the study including the follow up period.
* Any clinically significant medical condition (e.g., within six months of baseline, had myocardial infarction, angina pectoris, and/or congestive heart failure) that, in the opinion of the investigator, would compromise the safety of patient.
* Pulmonary Slow Vital Capacity (SVC) less than 65% of predicted for age, gender, and body type.
* Autoimmunity, including Crohn's disease or rheumatoid arthritis
* Current use of immunosuppressant medication or use of such medication within 4 weeks of Screening visit (Visit 1).
* Malignancy 5 years prior to enrollment, including melanoma,with the exception of localized skin cancers (with no evidence of metastasis, significant invasion, or re-occurrence within three years of baseline).
* Active systemic or local infection near the lumbar puncture site.
* Inability to lie flat for the duration of intrathecal cell transplantation, or inability to tolerate study procedures for any other reason.
* Other active systemic disease as defined by laboratory abnormalities delineated in Appendix IV.
* Use of herbal medications, nutritional supplements or other unapproved drugs or investigational medicinal products being used or studied for the treatment of ALS.
* Unwilling to forgo initiating the use of any new supplements during participation in the study.
* Enrolled in an investigational drug trial within 30 days of baseline visit
* Prior stem cell therapy for a neurological disease
* Kokmen Short Test of Mental Status score <32
* Presence of a tracheostomy
* Ventilator dependent
* Pregnancy
* Men or women of childbearing potential who are unwilling to employ adequate contraception
* Chronic low back pain requiring invasive procedures (i.e. epidural injections or lumbar spine surgery)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2017-10-10 (Actual); Primary Completion 2024-01-31 (Actual); Study Completion 2025-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Nathan P Staff, MD, PhD, Principal Investigator — Mayo Clinic; Anthony J Windebank, MD, Principal Investigator — Mayo Clinic
Locations (3):
- United States (3):
  - Mayo Clinic, Scottsdale, Arizona
  - Mayo Clinic, Jacksonville, Florida
  - Mayo Clinic in Rochester, Rochester, Minnesota

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 75 participants signed the informed consent form, however nine participants screened failed prior to being randomized.
Groups:
- Mesenchymal Stromal Cells: Autologous Adipose-derived Mesenchymal Stromal Cells (aaMSCs) were administered intrathecally at a single dose in a volume of 5-10 mL, all patients received 5 x 10^7 intrathecal aaMSCs at the first injection (Visit 4). Subsequent doses may be reduced to 1 x 10^7 or increased to 1 x 10^8, based on Dose Modification Rules.
  Autologous Adipose-derived Mesenchymal Stromal Cells: The investigational product consists of autologous adipose-derived Mesenchymal Stromal Cells (MSCs), suspended in 5-10 mL Lactated Ringer's. The MSC were provided in a sterile syringe labelled with appropriate patient and product identifiers ready for intrathecal injection.
Period: Overall Study
Arm/Group | Mesenchymal Stromal Cells
Started | 66
Completed | 57
Not Completed | 9
Not completed — Withdrawal by Subject | 6
Not completed — Physician Decision | 1
Not completed — Withdrawn due to disease progression | 2

BASELINE CHARACTERISTICS:
Arm/Group | Mesenchymal Stromal Cells
Number analyzed (Participants) | 57
Age, Continuous [Mean (Full Range); unit: years] | 56 [28 to 77]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 40
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 55
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 55
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 57

OUTCOME MEASURES:

1. Primary Outcome: Adverse Events
Description: The number of adverse events experienced by subjects
Time Frame: 12-months
Measure: Number; unit: Number of Adverse Events
Arm/Group | Mesenchymal Stromal Cells
Number analyzed (Participants) | 57
Number of Adverse Events | 668

2. Primary Outcome: Unexpected Severe Adverse Events
Description: The number of unexpected severe adverse events experienced by subjects
Time Frame: 12-months
Measure: Number; unit: Number of unexpected severe adverse eve
Arm/Group | Mesenchymal Stromal Cells
Number analyzed (Participants) | 57
Number of unexpected severe adverse eve | 41

3. Secondary Outcome: Change in Slope of ALS Functional Rating Scale - Revised (ALSFRS-R)
Description: The ALSFRS-R includes 12 questions. Each task is rated on a five-point scale from 0 = can't do, to 4 = normal ability. Individual item scores are summed to produce a reported score of between 0=worst and 48=best. The change in slope is the rate at which a patient's functional ability declines over time, as measured by the change in the ALFSFRS score over 1 year. A steeper slope signifies a faster decline in function. A negative change in slope indicates a decline in function and positive change in slope indicates an improvement in function.
Time Frame: baseline, approximately 1 year
Measure: Mean (Inter-Quartile Range); unit: Score on a scale/year
Arm/Group | Mesenchymal Stromal Cells
Number analyzed (Participants) | 57
Score on a scale/year | -0.11 [-1.19 to 0.93]
Statistical Analysis 1: Comparison: Mesenchymal Stromal Cells; Test type: Superiority; p = 0.38, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the time of enrollment through the end of the follow-up period, approximately 1 year.
Arm/Group | Mesenchymal Stromal Cells
All-Cause Mortality (participants affected / at risk) | 4/57
Serious Adverse Events (participants affected / at risk) | 26/57
Other Adverse Events (participants affected / at risk) | 56/57
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mesenchymal Stromal Cells (N=57)
Appendicitis (Infections and infestations) | 1 (1)
Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Disease Progression (General disorders) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 11 (11)
Fall (Injury, poisoning and procedural complications) | 1 (1)
Feeding Tube Placement (Gastrointestinal disorders) | 1 (1)
Fracture (Injury, poisoning and procedural complications) | 2 (2)
Gastrointestinal Disorders-Other (Gastrointestinal disorders) | 1 (1)
Hematoma (Vascular disorders) | 1 (1)
Infections and Infestations-Other (Infections and infestations) | 4 (5)
Intracranial Hemorrhage (Nervous system disorders) | 1 (1)
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 1 (2)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Stroke (Nervous system disorders) | 1 (1)
Superficial Thrombophlebitis (Vascular disorders) | 1 (1)
Upper Respiratory Infection (Infections and infestations) | 1 (1)
Weight Loss (Investigations) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mesenchymal Stromal Cells (N=57)
Back Pain (Musculoskeletal and connective tissue disorders) | 47 (101)
Headache (Nervous system disorders) | 33 (63)
Abdominal Pain (Gastrointestinal disorders) | 2 (2)
Abrasion on the left side of head (Injury, poisoning and procedural complications) | 1 (1)
Allergic Reaction (Immune system disorders) | 1 (1)
Anal Fissure (Gastrointestinal disorders) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1)
Arachnoiditis (Nervous system disorders) | 1 (1)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Bilateral Ankle Pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Bilateral Left Buttock Pain and Leg Pain Post Procedure (Musculoskeletal and connective tissue disorders) | 1 (1)
Black Hairy Tongue (Infections and infestations) | 1 (1)
Blood and Lymphatic System Disorders-Other (Blood and lymphatic system disorders) | 1 (1)
Bruising (Injury, poisoning and procedural complications) | 19 (41)
Buttock Pain (Musculoskeletal and connective tissue disorders) | 23 (33)
Chills (General disorders) | 1 (1)
Confusion (Psychiatric disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 10 (10)
Cough (Respiratory, thoracic and mediastinal disorders) | 6 (6)
Creatinine Increased (Investigations) | 1 (1)
Cystitis Noninfective (Renal and urinary disorders) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 3 (3)
Depression (Psychiatric disorders) | 3 (3)
Diarrhea (Gastrointestinal disorders) | 5 (6)
Dysarthria (Nervous system disorders) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 8 (8)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Face Edema (General disorders) | 1 (1)
Limb Edema (General disorders) | 4 (5)
Eye Disorder-Other (Eye disorders) | 3 (3)
Eye Infection (Infections and infestations) | 2 (2)
Facial Pain (General disorders) | 2 (2)
Fall (Injury, poisoning and procedural complications) | 44 (115)
Respiratory Fatigue (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Fecal incontinence (Gastrointestinal disorders) | 1 (1)
Feeding Tube Placement (Gastrointestinal disorders) | 1 (1)
Fever (General disorders) | 1 (2)
Food Poisoning (General disorders) | 1 (1)
Forehead Abrasion (Injury, poisoning and procedural complications) | 1 (1)
Fracture (Injury, poisoning and procedural complications) | 4 (4)
Gait Disturbance (General disorders) | 2 (2)
Gastroesophageal Reflux Disease (Gastrointestinal disorders) | 3 (3)
General Disorders and Administration Site Conditions-Other (General disorders) | 3 (7)
Hamstring Stiffness (Musculoskeletal and connective tissue disorders) | 1 (1)
Hangover Feeling (General disorders) | 1 (1)
Head Cold (Infections and infestations) | 4 (5)
Head Laceration (Injury, poisoning and procedural complications) | 1 (1)
Hematoma (Vascular disorders) | 1 (1)
Hemorrhoids (Gastrointestinal disorders) | 2 (2)
Hyperlipidemia (Metabolism and nutrition disorders) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1)
Hypotension (Vascular disorders) | 1 (1)
Infections and Infestations-Other (Infections and infestations) | 9 (9)
Influenza B (Infections and infestations) | 1 (1)
Ingrown Toe Nails (Skin and subcutaneous tissue disorders) | 2 (2)
Injection Site Soreness (General disorders) | 1 (1)
Injury, Poisoning and Procedural Complications-Other (Injury, poisoning and procedural complications) | 4 (6)
Laryngeal Inflammation (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Left Shoulder Abrasion (Injury, poisoning and procedural complications) | 1 (1)
Leg Pain (Musculoskeletal and connective tissue disorders) | 5 (5)
Low Back and Left Leg Pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Low Back Pain Tailbone (Musculoskeletal and connective tissue disorders) | 1 (1)
Low Back Pain and Upper Thigh Pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Lower Back Soreness (Musculoskeletal and connective tissue disorders) | 1 (1)
Lower Back Stiffness (Musculoskeletal and connective tissue disorders) | 1 (1)
Lung Infection (Infections and infestations) | 1 (1)
Muscle Cramp (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscle Weakness Lower Limb (Musculoskeletal and connective tissue disorders) | 2 (2)
Musculoskeletal and Connective Tissue Disorder-Other (Musculoskeletal and connective tissue disorders) | 3 (3)
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 9 (9)
Nausea (Gastrointestinal disorders) | 4 (4)
Neck Pain (Musculoskeletal and connective tissue disorders) | 6 (6)
Neoplasms Benign, Malignant and Unspecified (including cysts and polyps)-Other (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Norovirus Vomiting (Infections and infestations) | 1 (1)
Oral Thrush (Infections and infestations) | 2 (2)
Pain (General disorders) | 10 (21)
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 29 (65)
Pain of Skin (Skin and subcutaneous tissue disorders) | 2 (3)
Palpitations (Cardiac disorders) | 1 (1)
Paresthesia (Nervous system disorders) | 1 (1)
Post Injection Low Back and Left Leg Pain (Injury, poisoning and procedural complications) | 1 (1)
Postnasal Drip (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Productive Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Restlessness (Psychiatric disorders) | 1 (1)
Scabs on Face from Walking into a Cable (Injury, poisoning and procedural complications) | 1 (1)
Scalp Pain (Skin and subcutaneous tissue disorders) | 2 (2)
Sinus Infection (Infections and infestations) | 1 (1)
Sinus Tachycardia (Cardiac disorders) | 1 (1)
Sinusitis (Infections and infestations) | 2 (2)
Skin Ulceration (Skin and subcutaneous tissue disorders) | 3 (3)
Sore Throat (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Sore, Achy Hamstrings and Calves-Bilateral (Musculoskeletal and connective tissue disorders) | 1 (1)
Supraventricular Tachycardia (Cardiac disorders) | 1 (3)
Surgical and Medical Procedures-Other (Surgical and medical procedures) | 2 (3)
Swollen Feet (General disorders) | 1 (1)
Tailbone Pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 1 (1)
Upper Respiratory Infection (Infections and infestations) | 1 (1)
Urinary Frequency (Renal and urinary disorders) | 2 (2)
Urinary Retention (Renal and urinary disorders) | 1 (1)
Urinary Tract Infection (Infections and infestations) | 5 (10)
Urinary Urgency (Renal and urinary disorders) | 5 (5)
Vascular Access Complication (Injury, poisoning and procedural complications) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 4 (6)
Vomiting (Gastrointestinal disorders) | 4 (4)
Wrist Fracture (Injury, poisoning and procedural complications) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-12-19): https://cdn.clinicaltrials.gov/large-docs/03/NCT03268603/Prot_SAP_000.pdf